CLINICAL TRIAL: NCT01064193
Title: Influence of Local Biopsy of the Endometrium Prior to Controlled Ovarian Stimulation for IVF or ICSI Procedure on the Rates of Embryo Implantation, Clinical Pregnancy and Live Birth in ART
Brief Title: Impact of Local Biopsy to the Endometrium Prior to Controlled Ovarian Stimulation on Clinical Pregnancy
Acronym: NIDABRECHE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CHUBX 2009/12
Record Dates: First submitted 2010-02-05; First posted 2010-02-08 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Primary or Secondary Infertility
Keywords: In Vitro Fertilization; biopsy; pregnancy; Implantation; Embryo; first or second IVF tentative
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group 1 : IVF with biopsy (Experimental): fresh IVF-embryo transfer treated with long protocol or antagonist protocol for the controlled ovarian hyperstimulation plus local injury to the endometrium of patients one menstrual cycle before the IVF
  Interventions: Procedure: biopsy
- group 2 (Active Comparator): fresh IVF-embryo transfer treated with long protocol or antagonist protocol for the controlled ovarian hyperstimulation alone
  Interventions: Procedure: IVF

INTERVENTIONS:
Procedure: biopsy — The endometrium biopsy will be done as the same time as the GnRH treatment. The biopsy is realised with a Pipette de Cornier® (CDD international, PROMIDED France) following the laboratory protocol:
  * Apply antiseptic solution (povidone-iodine, Dakin®) on the cervix and vagina. In most cases, using Pozzi forceps is not necessary.
  * Insert carefully the pipelle de Cornier® in the uterus through the cervix.
  * Withdraw the piston to create a negative pression
  * Move the pipelle de cornier® in and out while twisting. Take care to no remove the pipelle form the uterus (suction lost). Twist the pipelle de Cornier® to cover an angle of 360°. Make several "in and out" cycle in order to collect a complete sample of the endometrium.
  * Withdraw the pipelle de Cornier® when filled with tissue
  * Reinsert internal piston to deposit sample in cup filled with a fixative.
  Arms: group 1 : IVF with biopsy
Procedure: IVF — fresh IVF-embryo transfer treated with long protocol for the controlled ovarian hyperstimulation
  Arms: group 2

SUMMARY:
In vitro fertilization (IVF) is the only available solution for many couples with various forms of infertility. The embryo implantation step in the IVF procedure is a complex multistage process and represents the majority of the causes of the IVF failure. Several approaches have been evaluated to improve implantation rates but none has demonstrated its superiority. However, endometrial receptivity is important for pregnancy and several studies suggest that local injury to the endometrium of IVF patients improves the rates of embryo implantation, clinical pregnancy and live birth.

DETAILED DESCRIPTION:
They are possible mechanisms by which endometrial sampling may increase receptivity and improve clinical pregnancy rate of IVF-ET. First, local injury to proliferative phase endometrium might induce the decidualization of the endometrium, and increase its implantation rate. Second, local injury to the endometrium might provoke the wound healing, involving a mass secretion of different cytokines and growth factor, which are beneficial for embryo implantation. Last, the injury might make the endometrium maturation.

This study proposes to evaluate the efficiency of an endometrial injury in the first controlled ovarian hyperstimulation cycle on the rate of clinical pregnancy, in assisted reproductive technologies. This study will compare 2 groups of patients. The first group will undergo biopsy of the endometrium before the IVF; the second will undergo the IVF alone. Inclusions will be conducted on 33 months; the patients will be in the study for a period of 36 weeks. The total duration of the study is 39 months

ELIGIBILITY:
Inclusion Criteria:

* primary or secondary infertility
* first or second IVF attempt
* aged ≥18 and ≤38 years
* regular menstrual cycles
* FSH≤ 12IU/L
* Informed consent signed

Exclusion Criteria:

* ovocyte donor
* pathology of the uterus or annexes
* Body mass index (BMI)> 35
* ongoing vaginal infection
* undetermined vaginal bleeding
* contraindication to the Cornier pipette or to these treatments : Gonal F®, Puregon®, Ovitrelle®, Utrogestan®,
* women included in another study on medically assisted procreation
* any administrative or legal supervision

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 190 (Actual)
Dates: Start 2010-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Rate of clinical pregnancy | 5 weeks after the embryo implantation in an IVF procedure

SECONDARY OUTCOMES:
Rate of clinical pregnancy | 3 months after the IVF implantation
Rate of embryo implantation | 5 weeks after the embryo implantation
Rate of miscarriage/extra-uterine pregnancy/multiple pregnancy | first trimester after the IVF
Adverse effects during the local injury (biopsy) to the endometrium | during the biopsy
Evaluation of the patients pain intensity and type from the biopsy. | during and after the biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Benard, Doctor, Study Chair — University Hospital Bordeaux, France; Sandrine Blancpain, Doctor, Principal Investigator — University Hospital Bordeaux, France
Locations (3):
- France (3):
  - CHU de Bordeaux, Hôpital Saint André, service de chirurgie gynécologie et médecine de la reproduction, Bordeaux
  - Cabinet Médical de gynécologie, Pessac
  - CHU de Toulouse, service de médecine et biologie de la reproduction, Toulouse

REFERENCES:
- [Background] Bourgain C, Devroey P. The endometrium in stimulated cycles for IVF. Hum Reprod Update. 2003 Nov-Dec;9(6):515-22. doi: 10.1093/humupd/dmg045. PMID 14714588
- [Background] Richter KS, Bugge KR, Bromer JG, Levy MJ. Relationship between endometrial thickness and embryo implantation, based on 1,294 cycles of in vitro fertilization with transfer of two blastocyst-stage embryos. Fertil Steril. 2007 Jan;87(1):53-9. doi: 10.1016/j.fertnstert.2006.05.064. Epub 2006 Nov 1. PMID 17081537
- [Background] Barash A, Dekel N, Fieldust S, Segal I, Schechtman E, Granot I. Local injury to the endometrium doubles the incidence of successful pregnancies in patients undergoing in vitro fertilization. Fertil Steril. 2003 Jun;79(6):1317-22. doi: 10.1016/s0015-0282(03)00345-5. PMID 12798877
- [Background] Raziel A, Schachter M, Strassburger D, Bern O, Ron-El R, Friedler S. Favorable influence of local injury to the endometrium in intracytoplasmic sperm injection patients with high-order implantation failure. Fertil Steril. 2007 Jan;87(1):198-201. doi: 10.1016/j.fertnstert.2006.05.062. PMID 17197286
- [Background] Pritts EA, Atwood AK. Luteal phase support in infertility treatment: a meta-analysis of the randomized trials. Hum Reprod. 2002 Sep;17(9):2287-99. doi: 10.1093/humrep/17.9.2287. PMID 12202415
- [Background] Revelli A, Dolfin E, Gennarelli G, Lantieri T, Massobrio M, Holte JG, Tur-Kaspa I. Low-dose acetylsalicylic acid plus prednisolone as an adjuvant treatment in IVF: a prospective, randomized study. Fertil Steril. 2008 Nov;90(5):1685-91. doi: 10.1016/j.fertnstert.2007.08.037. Epub 2007 Dec 11. PMID 18054934
- [Background] Khairy M, Banerjee K, El-Toukhy T, Coomarasamy A, Khalaf Y. Aspirin in women undergoing in vitro fertilization treatment: a systematic review and meta-analysis. Fertil Steril. 2007 Oct;88(4):822-31. doi: 10.1016/j.fertnstert.2006.12.080. Epub 2007 May 16. PMID 17509593
- [Background] Silver MM, Miles P, Rosa C. Comparison of Novak and Pipelle endometrial biopsy instruments. Obstet Gynecol. 1991 Nov;78(5 Pt 1):828-30. PMID 1923207
- [Background] Gellersen B, Brosens IA, Brosens JJ. Decidualization of the human endometrium: mechanisms, functions, and clinical perspectives. Semin Reprod Med. 2007 Nov;25(6):445-53. doi: 10.1055/s-2007-991042. PMID 17960529
- [Background] Lindhard A, Ravn V, Bentin-Ley U, Horn T, Bangsboell S, Rex S, Toft B, Soerensen S. Ultrasound characteristics and histological dating of the endometrium in a natural cycle in infertile women compared with fertile controls. Fertil Steril. 2006 Nov;86(5):1344-55. doi: 10.1016/j.fertnstert.2006.03.052. Epub 2006 Sep 14. PMID 16978615
- [Background] Homburg R, Pap H, Brandes M, Huirne J, Hompes P, Lambalk CB. Endometrial biopsy during induction of ovulation with clomiphene citrate in polycystic ovary syndrome. Gynecol Endocrinol. 2006 Sep;22(9):506-10. doi: 10.1080/09513590600921366. PMID 17071535
- [Background] Sulewski JM, Ward SP, McGaffic W. Endometrial biopsy during a cycle of conception. Fertil Steril. 1980 Dec;34(6):548-51. doi: 10.1016/s0015-0282(16)45193-9. PMID 7450073
- [Background] Wentz AC, Herbert CM 3rd, Maxson WS, Hill GA, Pittaway DE. Cycle of conception endometrial biopsy. Fertil Steril. 1986 Aug;46(2):196-9. doi: 10.1016/s0015-0282(16)49510-5. PMID 3732525
- [Background] Balasch J, Vanrell JA, Marquez M, Gonzalez-Merlo J. Endometrial biopsy inadvertently taken in the cycle of conception. Int J Gynaecol Obstet. 1984 Apr;22(2):95-9. doi: 10.1016/0020-7292(84)90020-1. PMID 6145645
- [Background] Giorgetti C, Terriou P, Auquier P, Hans E, Spach JL, Salzmann J, Roulier R. Embryo score to predict implantation after in-vitro fertilization: based on 957 single embryo transfers. Hum Reprod. 1995 Sep;10(9):2427-31. doi: 10.1093/oxfordjournals.humrep.a136312. PMID 8530679
- [Background] Abramov Y, Elchalal U, Schenker JG. Severe OHSS: An 'epidemic' of severe OHSS: a price we have to pay? Hum Reprod. 1999 Sep;14(9):2181-3. doi: 10.1093/humrep/14.9.2181. No abstract available. PMID 10469676
- [Background] Balasch J, Fabregues F, Arroyo V. Peripheral arterial vasodilation hypothesis: a new insight into the pathogenesis of ovarian hyperstimulation syndrome. Hum Reprod. 1998 Oct;13(1O):2718-30. doi: 10.1093/humrep/13.10.2718. PMID 9804220
- [Background] Govaerts I, Devreker F, Delbaere A, Revelard P, Englert Y. Short-term medical complications of 1500 oocyte retrievals for in vitro fertilization and embryo transfer. Eur J Obstet Gynecol Reprod Biol. 1998 Apr;77(2):239-43. doi: 10.1016/s0301-2115(97)00263-7. PMID 9578285
- [Background] Perrier D'hauterive S, Charlet-Renard C, Goffin F, Foidart M, Geenen V. [The implantation window]. J Gynecol Obstet Biol Reprod (Paris). 2002 Sep;31(5):440-55. French. PMID 12379828
- [Background] Bourgain C. [Endometrial biopsy in the evaluation of endometrial receptivity]. J Gynecol Obstet Biol Reprod (Paris). 2004 Feb;33(1 Pt 2):S13-7. doi: 10.1016/s0368-2315(04)96397-1. French. PMID 14968038
- [Background] Zhou L, Li R, Wang R, Huang HX, Zhong K. Local injury to the endometrium in controlled ovarian hyperstimulation cycles improves implantation rates. Fertil Steril. 2008 May;89(5):1166-1176. doi: 10.1016/j.fertnstert.2007.05.064. Epub 2007 Aug 6. PMID 17681303
- [Background] Cornier E. The Pipelle: a disposable device for endometrial biopsy. Am J Obstet Gynecol. 1984 Jan 1;148(1):109-10. doi: 10.1016/s0002-9378(84)80043-5. No abstract available. PMID 6691367
- [Background] Check JH, Chase JS, Nowroozi K, Wu CH, Chern R. Clinical evaluation of the Pipelle endometrial suction curette for timed endometrial biopsies. J Reprod Med. 1989 Mar;34(3):218-20. PMID 2724236
- [Background] Henig I, Chan P, Tredway DR, Maw GM, Gullett AJ, Cheatwood M. Evaluation of the Pipelle curette for endometrial biopsy. J Reprod Med. 1989 Oct;34(10):786-9. PMID 2795561
- [Background] Machado F, Moreno J, Carazo M, Leon J, Fiol G, Serna R. Accuracy of endometrial biopsy with the Cornier pipelle for diagnosis of endometrial cancer and atypical hyperplasia. Eur J Gynaecol Oncol. 2003;24(3-4):279-81. PMID 12807240
- [Background] Golan A, Ron-el R, Herman A, Soffer Y, Weinraub Z, Caspi E. Ovarian hyperstimulation syndrome: an update review. Obstet Gynecol Surv. 1989 Jun;44(6):430-40. doi: 10.1097/00006254-198906000-00004. No abstract available. PMID 2660037
- [Derived] Frantz S, Parinaud J, Kret M, Rocher-Escriva G, Papaxanthos-Roche A, Creux H, Chansel-Debordeaux L, Benard A, Hocke C. Decrease in pregnancy rate after endometrial scratch in women undergoing a first or second in vitro fertilization. A multicenter randomized controlled trial. Hum Reprod. 2019 Jan 1;34(1):92-99. doi: 10.1093/humrep/dey334. PMID 30496529